CLINICAL TRIAL: NCT04761159
Title: Effect of Ketamin+Propofol Mixture on Postoperative Recovery
Brief Title: Ketamin Plus Propofol for Anesthesia Induction
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, ebru biricik, associate professor, Cukurova University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Ketamin-propofol
Record Dates: First submitted 2021-01-28; First posted 2021-02-18 (Actual); Last update posted 2023-04-20 (Actual); Status verified 2022-01

CONDITIONS: Postoperative Recovery
MeSH Terms: interventions — Ketamine

STUDY DESIGN:
Intervention Model Description: Randomised, controlled
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Ketofol1/1 (Active Comparator): Propofol 1 mg/kg + ketamin1 mg/kg (1/1 ratio) for group I to anesthesia induction.
  Interventions: Drug: Ketamine
- Ketofol1/2 (Active Comparator): propofol 1,5 mg/kg + ketamin 0,75 mg/kg (2/1 ratio) for group II to anesthesia induction
  Interventions: Drug: Ketamine
- Ketofol1/3 (Active Comparator): propofol 2 mg/kg +ketamin 0,66 mg/kg (3/1 ratio) for group III to anesthesia induction
  Interventions: Drug: Ketamine
- propofol (Active Comparator): propofol 3 mg/kg will perform for anesthesia induction
  Interventions: Drug: Ketamine

INTERVENTIONS:
Drug: Ketamine — Different mixture of ketamin-propofol will apply for anesthesia induction.
  Other Names: ketofol

SUMMARY:
ASA I-II 112 pediatric patients will recruit who underwent adenoidectomy-tonsillectomy surgery. Propofol 1 mg/kg + ketamin1 mg/kg (1/1 ratio) for group I; propofol 1,5 mg/kg + ketamin 0,75 mg/kg (2/1 ratio) for group II; propofol 2 mg/kg +ketamin 0,66 mg/kg (3/1 ratio) for group III; propofol 3 mg/kg will perform for anesthesia induction. General anesthesia will maintenance with sevoflurane 1-2% and O2/N2O mixture. Morphine 0.1mg/kg IV will be apply for postoperative analgesia at 10 min of anesthesia. Extubation time, length of stay in PACU, Watcha score, FLACC score will record. Than all data will statistically analyse.

DETAILED DESCRIPTION:
ASA I-II 112 pediatric patients will recruit who underwent adenoidectomy-tonsillectomy surgery in this randomised controlled study. The participants will divide into the 4 groups with computered random generation. The Different combination of propofol+ketamin mixture will apply at the induction of anesthesia. The groups will assign as group I,II, III and IV. Propofol 1 mg/kg + ketamin1 mg/kg (1/1 ratio) for group I; propofol 1,5 mg/kg + ketamin 0,75 mg/kg (2/1 ratio) for group II; propofol 2 mg/kg +ketamin 0,66 mg/kg (3/1 ratio) for group III; propofol 3 mg/kg will perform for anesthesia induction. Fentanyl 1 microgram per kg and rocuronium 0.6 mg/kg will apply for anesthesia induction to the all participants. General anesthesia will maintenance with sevoflurane 1-2% and O2/N2O mixture. Morphine 0.1mg/kg IV will be apply for postoperative analgesia at 10 min of anesthesia. Extubation time, length of stay in PACU, Watcha score, FLACC score will record. Than all data will statistically analyse.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II patients
* Underwent adenoidectomy-tonsillectomy surgery
* Age between 3-12

Exclusion Criteria:

* ASA III-IV patients
* Age; under 3 years old
* Age; above 12 years old.

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 112 (Actual)
Dates: Start 2021-02-15 (Actual); Primary Completion 2022-12-15 (Actual); Study Completion 2022-12-15 (Actual)

PRIMARY OUTCOMES:
Delirium score | 30 minutes in PACU
  Watcha scores will record till the patient discharge from the PACU.

SECONDARY OUTCOMES:
length of stay in PACU | 30 minutes in PACU
  The participants will observe in PACU till the Aldrete score will achieve 15. This duration of time will record.

CONTACTS AND LOCATIONS:
Locations (1):
- Cukurova University, Adana, Turkey (Türkiye)